CLINICAL TRIAL: NCT04757090
Title: A Pilot Study of 89Zr-Trastuzumab PET/CT in Subjects With Previously Treated HER2-Positive Solid Tumors Scheduled to Receive Treatment With MT-5111
Brief Title: 89Zr-Trastuzumab PET/CT in Subjects With Previously Treated HER2-Positive Solid Tumors Scheduled to Receive Treatment With MT-5111
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient staff
Sponsor: Washington University School of Medicine (Other)
Collaborators: Molecular Templates, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202103039
Record Dates: First submitted 2021-02-15; First posted 2021-02-16 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: HER2-positive Solid Tumor; HER-2 Positive Cancer
MeSH Terms: interventions — zirconium-89-trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 89Zr-trastuzumab PET/CT imaging (Experimental): * Enrolled subjects will be asked to undergo 18F-FDG PET/CT imaging (if not performed within the previous 90 days) and 89Zr-trastuzumab PET/CT imaging at baseline prior to the start of monotherapy MT-5111 treatment. Standard of care 18F-FDG PET/CT examinations performed within 90 days of 89Zr-trastuzumab administration can be used in place of a study specific 18F-FDG PET/CT scan. Baseline 89Zr-trastuzumab imaging should be completed no more than 30 days prior to initiating treatment with MT-5111.
  * Cold trastuzumab and 89Zr-trastuzumab will be administered at Visit 1 and the 89Zr-trastuzumab PET/CT (Visit 2) will take place 4 days (+/-1 day) after administration of 89Zr-trastuzumab.
  Interventions: Drug: 89Zr-trastuzumab

INTERVENTIONS:
Drug: 89Zr-trastuzumab — -To minimize uptake of the 89Zr-trastuzumab in normal tissues, immediately prior to planned 89Zr-trastuzumab injection patients will receive a 50 mg dose of "cold" unlabeled trastuzumab intravenously (IV). The administration of a fixed small dose of unlabeled antibody to improve tumor-to-normal-tissue (T/N) uptake of the radiolabeled antibody is standard in this type of imaging procedure.

SUMMARY:
This is an open-label, single center, pilot study to assess the feasibility of baseline 89Zr-trastuzumab PET/CT to predict response to treatment with monotherapy MT-5111

ELIGIBILITY:
Inclusion Criteria:

* Must meet eligibility criteria and be registered to receive treatment under Protocol MT-5111_001 (WU HRPO # 201907092).
* Must have at least one measurable lesion by RECIST 1.1 during the dose expansion phase of MT-5111_001. Osteosarcoma subjects with evaluable (e.g., bone-only) disease may be included.
* Must have standard of care 18F-FDG-PET/CT within 90 days before administration of 89Zr-trastuzumab OR be willing to undergo 18F-FDG PET/CT scan for research purposes.
* Able to undergo PET/CT imaging
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Hepatic only disease
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Average 89Zr-trastuzumab SUVmax of lesions identified on baseline FDG-PET/CT | At baseline
  -SUVmax is maximum standardized uptake value

SECONDARY OUTCOMES:
Average 89Zr-trastuzumab tumor-to-normal tissue uptake ratio of lesions identified on baseline FDG-PET/CT | At baseline
Average 89Zr-trastuzumab tumor-to-blood uptake ratio of lesions identified on baseline FDG-PET/CT | At baseline
Intra-patient 89Zr-trastuzumab tumor uptake heterogeneity in patients with multiple lesions (fractions of scan-positive and scan-negative lesions) | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Van Tine, M.D., Ph.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu